CLINICAL TRIAL: NCT06020209
Title: Cardiac Computed Tomography for Comprehensive Risk Stratification of Arrhythmic, Atherothrombotic and Heart Failure Events Following Reperfused ST-segment Elevation Myocardial Infarction
Brief Title: CCT for Comprehensive Risk Stratification Following STEMI
Acronym: CT-STEMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: A.O.U. Città della Salute e della Scienza - Molinette Hospital (Other); Istituto Auxologico Italiano (Other); University of Messina (Other); Ministry of Health, Italy (Other Government)
Responsible Party: Principal Investigator, Marco Gatti, Principal Investigator, University of Turin, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CT-STEMI; GR-2021-12372092 (Other Grant/Funding Number: Ministry of Health, Italy)
Record Dates: First submitted 2023-07-13; First posted 2023-08-31 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Myocardial Infarction
Keywords: ST Elevation Myocardial Infarction; Coronary Artery Disease; Computed Tomography (CT); Cardiovascular Magnetic Resonance (CMR); Risk assessment
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STEMI patients (Experimental): Patients with reperfused ST-segment Elevation Myocardial Infarction
  Interventions: Diagnostic Test: Cardiac Computed Tomography; Diagnostic Test: Cardiac Magnetic Resonance

INTERVENTIONS:
Diagnostic Test: Cardiac Computed Tomography — A comprehensive CCT protocol will be performed in the post-acute phase of STEMI. Specifically, the CCT protocol will include a pre-contrast scan and an angiographic scan ( also set up to assess ventricular volume and function) followed by late contrast enhancement scan.
Diagnostic Test: Cardiac Magnetic Resonance — A comprehensive CMR protocol will be performed in the post-acute phase of STEMI. Specifically, the CMR protocol is designed for morpho-functional analysis and tissue characterisation (including assessment of late gadolinium enhancement and mapping). CMR will be considered the gold standard.

SUMMARY:
The CT-STEMI study aims to evaluate a comprehensive cardiac computed tomography (CCT) protocol for assessing the risk of heart failure (HF), life-threatening arrhythmias (LTA), and atherothrombotic events following ST-elevation myocardial infarction (STEMI). This multicenter, prospective study has three main objectives:

1. Comparing the diagnostic accuracy of the comprehensive CCT protocol with cardiac magnetic resonance (CMR), considered the non-invasive gold standard.
2. Determining the prognostic value of CCT in assessing myocardial tissue adverse features related to STEMI.
3. Evaluating the atherosclerotic burden in patients with post-acute STEMI.

Two hundred patients will undergo both CCT and CMR in the post-acute phase, and their follow-up will focus on monitoring HF, LTA, and ischemic events. The CT-STEMI study represents the first attempt to assess the potential of CCT in providing a comprehensive risk assessment following STEMI in a large contemporary population. The findings of this study have the potential to revolutionize post-STEMI risk stratification practices.

DETAILED DESCRIPTION:
Background / State of Art

STEMI remains a leading cause of mortality. In the first year, STEMI survivors face an incident burden of heart failure (HF) as high as 25%, of ischemic events up to 18.3% and of LTA up to 1.5%.

CMR has emerged as the most potent tool to predict adverse left ventricular (LV) remodeling following STEMI. Infarct size (IS), microvascular obstruction (MVO) and intramyocardial hemorrhage (IMH) measured by CMR are all independent HF predictors, able to outperform clinical and reperfusion parameters and to predict long-term adverse remodeling among patients with initially preserved LV ejection fraction (LVEF).

Systematic CMR implementation following STEMI into routine clinical practice is difficult for several reasons, including limited availability, high costs as well as practical issues such as time and staff allocation. Moreover, CMR does not assess the coronary tree failing to provide a risk assessment comprehensive of the atherothrombotic component, beyond HF and arrhythmias.

Since recent advances in CCT technology have expanded its applicability beyond accurate morpho-functional assessment to the characterization of the myocardium, allowing for quantification of IS, MVO and extracellular volume (ECV). CCT may now offer unprecedent opportunities to provide a comprehensive risk assessment following STEMI with an ever-increasing available technology, with moderate costs and logistic effectiveness, and with very low radiation dose exposure with current scanners and protocols.

Hypotesis and Significance

Despite giant leaps forward in the acute and chronic management, STEMI remains a leading cause of mortality and morbidity worldwide.

Risk stratification is the foundation to tailoring treatment selection and intensity. However, the current tools to predict adverse events following STEMI including HF development, recurrent atherothrombotic events and life-threatening arrhythmias have poor prediction abilities or require cumbersome and often unavailable diagnostic technologies.

CMR has emerged as the most potent tool to predict adverse LV) remodeling following STEMI. Current post-MI arrhythmic risk stratification to mandate implantable cardioverter defibrillator implantation is chiefly based on LV EF. However, the evaluation of scar burden by CMR may outperform EF to predict life-threatening arrhythmias and has the potential to improve management among patients without a current indication for an implantable cardioverter defibrillator.

Systematic CMR implementation following STEMI into routine clinical practice is difficult for several reasons, including limited availability, high costs as well as practical issues such as time and staff allocation. Moreover, while providing excellent myocardial tissue characterization, CMR does not assess the coronary tree failing to provide a risk assessment comprehensive of the atherothrombotic component, beyond HF and arrhythmias.

Since recent advances in CCT technology have expanded its applicability beyond accurate morpho-functional assessment to the characterization of the myocardium, CCT may now offer unprecedent opportunities to provide a comprehensive risk assessment following STEMI with an ever-increasing available technology, with moderate costs and logistic effectiveness, and with very low radiation dose exposure with current scanners and protocols.

While preliminary data on the CCT performance to assess myocardial tissue characteristics are promising, accurate validation of this technology against CMR and clinical outcomes in large populations will be pivotal for clinical implementation. Moreover, the application of this technology to stratify HF and arrhythmic risk following STEMI has never been assessed.

The CT-STEMI study will be the first to assess the potential of CCT to provide a comprehensive risk assessment following STEMI in a large contemporary population, to lay the bases for a paradigm shift in post-STEMI risk stratification.

Specific Aim 1 To compare the diagnostic accuracy of a comprehensive CCT protocol to that of CMR, the non-invasive gold standard.

Specific Aim 2 To determine the prognostic value of CCT-assessed myocardial tissue STEMI-related adverse features.

Specific Aim 3 To evaluate the atherosclerotic burden in patients with post-acute STEMI.

For this purpose, in this prospective study, a total of two hundred patients will be recruited and undergo coronary computed tomography (CCT) and cardiac magnetic resonance imaging (CMR) during the post-acute phase of ST-elevation myocardial infarction (STEMI).

Experimental Design Aim 1

The CMR study will be used as the reference standard to assess the accuracy of CCT in evaluating morpho-functional parameters such as Left Ventricular End-Diastolic Volume (LVEDV), Left Ventricular End-Systolic Volume (LVESV), LVEF, Right Ventricular End-Diastolic Volume (RVEDV), Right Ventricular End-Systolic Volume (RVESV), and Right Ventricular Ejection Fraction (RVEF). Additionally, the study will also examine myocardial tissue characteristics including IS, myocardial edema, MVO, IMH, and ECV.

Experimental Design Aim 2

The patients will undergo follow-up procedures starting from the commencement of the study. Co-primary endpoints will be:

* Atherothrombotic primary endpoint: composite of recurrent acute coronary syndrome, ischemic stroke or cardiovascular death
* HF and arrhythmic primary endpoint: composite of new congestive HF or sustained ventricular arrhythmia or appropriate Implantable Cardioverter-Defibrillator (ICD) intervention or sudden cardiac death or resuscitated cardiac arrest

Individual CCT predictors (EF, IS, myocardial edema, MVO, IMH and ECV) will be evaluated and compared with those derived from CMR.

Experimental Design Aim 3

The purpose of this sub-study is to report the prevalence and features of non-culprit plaques, as well as to investigate the independent predictive significance of CCT-assessed coronary plaque characteristics on event prediction.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* STEMI diagnosis
* Primary Percutaneous Coronary Intervention (PCI) <24h from symptom onset
* Hemodynamic stability without inotropic support within 4 days from the index event

Exclusion Criteria:

* Known chronic kidney disease with estimated Glomerular Filtration Rate (GFR) < 30 mL/min/1.73mq
* History of allergic reaction to CCT or CMR contrast media
* Inability or unwilling to undergo CCT or CMR scanning
* Pregnancy or breast-feeding
* Severe atrial or ventricular arrhythmia burden
* Severe valvular stenosis or regurgitation
* Prior clinical congestive HF diagnosis (asymptomatic LV dysfunction can be included)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
CCT - diagnostic accuracy | Baseline
  CMR study will be used as the reference standard to assess the accuracy of CCT in evaluating morpho-functional parameters such as
  * LVEDV (ml)
  * LVESV (ml)
  * LVEF (%)
  * RVEDV (ml)
  * RVESV (ml)
  * RVEF (%)
  Additionally, the study will also examine myocardial tissue characteristics including:
  * IS: presence or absence
  * IS (gr)
  * IS (% of the total left ventricular mass)
  * Myocardial edema: presence or absence
  * Myocardial edema (gr)
  * Myocardial edema (% of the total left ventricular mass)
  * MVO: presence or absence
  * MVO (gr)
  * MVO (% of the total left ventricular mass)
  * IMH: presence or absence
  * IMH (gr)
  * IMH (% of the total left ventricular mass)
  * ECV (%)
CCT - risk stratification | 1 month, 1 year
  Individual CCT predictors will be evaluated and compared with those derived from CMR:
  * IS: presence or absence
  * IS (gr)
  * IS (% of the total left ventricular mass)
  * Myocardial edema: presence or absence
  * Myocardial edema (gr)
  * Myocardial edema (% of the total left ventricular mass)
  * MVO: presence or absence
  * MVO (gr)
  * MVO (% of the total left ventricular mass)
  * IMH: presence or absence
  * IMH (gr)
  * IMH (% of the total left ventricular mass)
  * ECV (%)
CCT - Coronary artery disease (CAD) impact of risk stratification | Baseline, 1 month, 1 year
  CCT Report include prevalence and features of non-culprit plaques with a qualitative analysis, based on the presence of:
  * positive remodeling: presence or absence
  * low attenuation plaque: presence or absence
  * spotty calcification: presence or absence
  * "napkin ring" sign: presence or absence
  and semi-quantitative analysis with a dedicated cardiac CT software:
  * Plaque burden (%)
  * Plaque volume (per lesion and per vessel) (mm^3)
  * Vessel remodeling index (ratio)
  * Mean plaque and lumen intensities (HU)
  * Plaque characterization components: presence or absence of Dense Calcium, Necrotic Core, Fibrous Fatty, Fibrous
  * Evaluation of Peri Vascular Adipose Tissue (PVAT) - thickness measurement in millimeters (mm)
  * Evaluation of Peri Vascular Adipose Tissue (PVAT) - volume measurement in millimeters cubed (mm^3)
  Finally this data will used to investigate the independent predictive significance of CCT-assessed coronary plaque characteristics on event prediction.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Gatti, M.D., Principal Investigator — University of Turin, Italy
Locations (3):
- Italy (3):
  - Azienda Ospedaliera Policlinico Universitario "G. Martino", Messina
  - Istituto Auxologico Italiano - IRCCS - Ospedale San Luca, Milan
  - A.O.U. Città della Salute e della Scienza - Molinette Hospital, Turin

IPD SHARING:
Plan to Share IPD: No